CLINICAL TRIAL: NCT02065076
Title: Efficacy of Sodium Polystyrene Sulfonate in the Treatment of Hyperkaliemia in Ambulatory Pre-dialysis Outpatients : a Randomized Triple-blind Placebo-controlled Trial
Brief Title: Efficacy of Sodium Polystyrene Sulfonate in the Treatment of Hyperkaliemia in Pre-dialysis Patients
Acronym: SKIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Principal Investigator, Dr. Vincent Pichette, M.D., Ph.D., FRCP(C), nephrologist, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13089
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Hyperkalemia; Chronic Kidney Failure
Keywords: Sodium Polystyrene Sulfonate; Kayexalate; Pre-dialysis; Outpatients; Hyperkalemia; Chronic kidney failure; Potassium
MeSH Terms: conditions — Hyperkalemia; Kidney Failure, Chronic | interventions — polystyrene sulfonic acid; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium Polystyrene Sulfonate (Active Comparator): 30 g sodium polystyrene sulfonate powder, mixed with water qs ad 150 ml, taken PO once daily for seven days
  Interventions: Drug: Sodium polystyrene sulfonate
- Lactose with carob gum (Placebo Comparator): 30 g placebo powder, mixed with water qs ad 150 ml, taken PO once daily for seven days
  Interventions: Drug: Lactose with carob gum

INTERVENTIONS:
Drug: Sodium polystyrene sulfonate
  Other Names: SPS; Kayexalate; Solystat
  Arms: Sodium Polystyrene Sulfonate
Drug: Lactose with carob gum
  Other Names: Placebo
  Arms: Lactose with carob gum

SUMMARY:
The purpose of this trial is to determine if sodium polystyrene sulfonate (SPS) is an effective treatment of mild hyperkalemia in chronic kidney disease patients followed at a pre-dialysis or nephrology outpatient clinic. Subjects will be randomized to one of two treatment arms: 30 g of placebo or SPS to be taken orally once daily for seven days. The change in serum potassium levels will be compared in both treatment groups. The proportion of subjects attaining normokalemia (3.5 to 5.0 mmol/L) after seven days of treatment will also be compared. Finally, side effects will be reported for each treatment arm.

DETAILED DESCRIPTION:
Background

Hyperkalemia affects up to 10% of patients suffering from chronic kidney failure and up to 42% of patients with an estimated glomerular filtration rate lower than 20 mL/min/1.73m2. There is currently limited evidence on the use of sodium polystyrene sulfonate for the treatment of mild hyperkalemia. There are even fewer trials supporting its use over several days. To our knowledge, only one other study has evaluated its chronic use in fourteen patients, but hadn't controlled for recent changes in medications. Since its use is associated with adverse events that can considerably affect patients' quality of life, it appears primordial to better assess its place in the treatment of hyperkalemia in pre-dialysis patients.

Methods

The aim of this trial is to evaluate the use of sodium polystyrene sulfonate in the treatment of mild asymptomatic hyperkalemia in predialysis patients. Participants will be randomized to receive either 30 g of placebo or 30 g of SPS orally once daily for seven days. Serum potassium levels will be assessed at baseline and on the day following the last dose of their treatment. The change in serum potassium levels and the proportion of patients attaining normokalemia will be compared between study groups. The incidence of adverse events (nausea, diarrhea, constipation, electrolyte disorders) will also be reported. Participants will also be asked to fill out a food diary for 3 out of the 7 study days. This diary will be used to estimate each participant's average daily intake of potassium and therefore evaluate the similarity of diets between both intervention arms.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over
* Outpatients followed at the pre-dialysis or nephrology clinics of Maisonneuve-Rosemont Hospital
* Subjects who have taken SPS in the past 7 days: serum potassium level measured for their regular followup of 4.5 to 5.5 mmol/L, inclusive, and serum potassium level of 5.0 to 5.9 mmol/L, inclusive, after a one week washout period
* Subjects who have not taken SPS in the past 7 days: serum potassium levels measured for their regular followup and on the day of randomisation of 5.0 to 5.9, inclusive

Exclusion Criteria:

* Subjects with a contraindication to SPS : known hypersensitivity to the product, history of obstructive bowel disease, patients at high risk of obstructive bowel disease
* Subjects unable of giving informed consent
* Subjects with severe or symptomatic hyperkalemia requiring a treatment
* Subjects on dialysis (hemodialysis or peritoneal dialysis)
* Women who are pregnant or breastfeeding
* Subjects who have had a change in the dosage of insulin in the past week, if this change represents more than 10% of the daily total dose or more than 5 units
* Subjects who stopped, started or changed the dosage of an angiotensin converting enzyme inhibitor, an angiotensin II receptor blocker or aliskiren in the past 60 days
* Subjects who stopped, started or changed the dosage of another medication affecting serum potassium levels in the past 30 days
* Subjects who have had an episode of decompensated heart failure in the past 30 days
* Subjects currently enrolled on another research protocol
* Subjects who are lactose intolerant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in serum potassium levels from baseline | After 7 days
  Compare the change in serum potassium levels from baseline in both treatment arms after 7 days of treatment with SPS or placebo 30 g once daily

SECONDARY OUTCOMES:
Proportion of subjects attaining normokalemia (serum potassium level of 3.5 to 5.0 mmol/L) in each treatment arm | After 7 days
  Compare the proportion of subjects attaining normokalemia (serum potassium level of 3.5 to 5.0 mmol/L) in each arm after one week of sodium polystyrene sulfonate or placebo
Number of patients with adverse events in each treatment group | Up to 7 days
  Report the number of patients with adverse events, notably nausea, diarrhea, constipation, electrolyte disorders (hypomagnesemia, hypernatremia, hypophosphatemia, hypocalcemia, hypokalemia)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Pichette, MD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Saglimbene VM, Strippoli GF. Potassium binders for chronic hyperkalaemia in people with chronic kidney disease. Cochrane Database Syst Rev. 2020 Jun 26;6(6):CD013165. doi: 10.1002/14651858.CD013165.pub2. PMID 32588430